CLINICAL TRIAL: NCT01113333
Title: A Double Blind, Placebo Controlled Ascending Single Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of the IKK Inhibitor, SAR113945, Following Intra-articular Administration in Patients With Knee Osteoarthritis
Brief Title: Safety, Tolerability and Pharmacokinetics of SAR113945 Following Intra-articular Administration in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDU10820; 2009-017502-36 (EudraCT Number); U1111-1116-5630 (Other: UTN)
Record Dates: First submitted 2010-04-23; First posted 2010-04-29 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAR113945 (Experimental): SAR113945, single dose according to dose escalation design
  Interventions: Drug: SAR113945
- Placebo (Placebo Comparator): 0.9% saline solution, single dose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Pharmaceutical form:injection
  Route of administration: intra-articular
  Arms: Placebo
Drug: SAR113945 — Pharmaceutical form:injection
  Route of administration: intra-articular
  Arms: SAR113945

SUMMARY:
Primary Objective:

* Assess the safety and tolerability of single intra-articular doses of SAR113945 in patients with knee osteoarthritis.

Secondary Objective:

* Assess systemic exposure of SAR113945 following intra-articular delivery.

DETAILED DESCRIPTION:
The total study duration per subject ranges from 4 to 20 weeks broken down as follows:

* screening within 4 weeks before dosing,
* follow-up of 4 weeks (28 days) after the single dose of study medication,
* prolonged by a maximum of 12 weeks if plasma PK level > Limit Of Quantification (LOQ) at Day 28.

ELIGIBILITY:
Inclusion criteria:

* Male patients or female patients of non child-bearing potential, aged at least 40 years with primary knee osteoarthritis having:

  * X-ray or Magnetic Resonance Imaging (MRI) evidence for Kellgren Lawrence Grades II./III joint space narrowing and osteophyte formation,
  * Western Ontario MacMaster (WOMAC) score ≦ 72,
  * American College of Rheumatology (ACR) Clinical and Radiographic criteria for osteoarthritis.

Exclusion criteria:

* Any uncontrolled, chronic condition or laboratory finding which, in the opinion of the Principal Investigator, could potentially put the patient at increased risk.
* Secondary osteoarthritis.
* Moderate/severe renal impairment.
* Underlying hepatobiliary disease and/or elevated Alanine Aminotransferase (ALT) > 3 Upper Limit of Normal range.
* Intra-articular injection within 3 months.
* Presence of local skin abnormality at the affected knee joint.
* Unable to be maintained for at least 2 weeks prior to entry into study on paracetamol or metamizole as analgesic.
* Any Investigational Product within 3 months.
* Any patient unlikely to comply with the requirements of the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Standard safety investigations (Physical examinations, 12 lead ECGs, vital signs (Blood pressure, heart rate, body temperature) and laboratory tests (hematology/coagulation, biochemistry, quantitative urinalysis)) | 4 weeks up to a maximum of 12 weeks
Examination of skin/soft tissue of injected knee | 4 weeks up to a maximum of 12 weeks
  Any reaction is classified as erythema, oedema, pain, papulae, haematoma and graded none, mild, moderate or severe.
Examination of knee joint of injected knee | 4 weeks up to a maximum of 12 weeks
  Any reaction is classified as effusion/worsening of effusion, warm and pain.

SECONDARY OUTCOMES:
Pharmacokinetic parameters for SAR113945 and potential metabolites(s) from plasma concentration (i.e. AUC, Cmax, tmax, t1/2) | 4 weeks up to a maximum of 16 weeks
Pharmacodynamic parameters (WOMAC Index, biomarkers relating to inflammation and cartilage/bone turnover) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Investigational Site Number 276001, Berlin, Germany